CLINICAL TRIAL: NCT04068025
Title: The Effect of Information, Motivation, Behavioral Skills Model on Urinary Incontinence and Quality of Life in Men With Overactive Bladder: A Randomized Controlled Trial
Brief Title: Information, Motivation, Behavioral Skills Model on Urinary Incontinence and Quality of Life in Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 16.01.2018 18/10
Record Dates: First submitted 2019-06-22; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Overactive Bladder; Quality of Life
Keywords: incontinence; male; overactive bladder; quality of life
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention: Control group (No Intervention): Patients in the control group were given usual care by a health professional who was not involved in the study and who worked in the Department of Urology. After the end of the study, the patients in the control group were also given structured bladder training similar to the patients in the intervention group.
- the IMB model (Active Comparator): Structured bladder training was applied to the patients in the intervention group via the IMB model.
  Interventions: Other: Assigned Interventions

INTERVENTIONS:
Other: Assigned Interventions — Information: In the information step of the bladder training program given through the IMB model, training was given about pelvic floor muscle exercises, bladder program formation, and lifestyle change. The training was conducted face-to-face by the nurse researcher for about 15-20 min, and the training booklet was given to the patients.
  Motivation: The patients in the intervention group were interviewed by the nurse researcher by phone or face-to-face in the 1st, 3rd, and 6th months after the training. The patients were motivated by providing information and counseling on the necessary issues. This process was carried out using motivational interviewing principles. Patients were given positive behavioral feedback and encouraged to control urinary incontinence.
  Behavioral Skills: Behavioral skills related to urinary incontinence were evaluated 6 months after the training,together with their effects on urinary incontinence symptom score and quality of life.
  Arms: the IMB model

SUMMARY:
Multiple studies have shown that education based on the IMB model is effective at bringing about health-related behavior change. The IMB model was found to be effective in developing healthy behaviors aimed at maintaining heart health, providing behavior to prevent smoking addiction, diabetes management, correct nutrition in iron deficiency anemia, and using condoms to prevent HIV. There are no studies in the literature regarding the adaptation of the IMB model to behavioral therapy in patients with OAB or urinary incontinence. To address this, there we aimed to investigate the effect of the IMB model on urinary incontinence and quality of life in men with OAB.

DETAILED DESCRIPTION:
This study aimed to investigate the effect of the Information, Motivation, Behavioral Skills Model (IMB) on urinary incontinence and quality of life in men with overactive bladder.

This is a single-center, parallel-group, open-label, randomized controlled clinical trial.

This study was conducted between February 2018 and February 2019, with a total of 60 male patients admitted to the urology clinic of a training and research hospital. Patients over the age of 18, male, and with overactive bladder were included in the study.

Participants were randomized into two equal groups: the intervention group (n=30) and control group (n=30). Structured bladder training with the IMB model was applied to the intervention group. This model was not applied to the control group. The primary outcome was the mean score change over the severity of incontinence measured by the International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF). The other outcomes were measured by the Urogenital Distress Inventory (UDI-6), Incontinence Impact Questionnaire-7 (IIQ-7), and Urinary Incontinence Information Rating scores. All outcome measures were evaluated before and 6 months after the training. Bladder training with IMB model was found to be effective at ameliorating urinary incontinence and improving quality of life in patients with an overactive bladder.

ELIGIBILITY:
Inclusion Criteria:

* Male patient
* Over 18 years old
* Overactive Bladder
* Urge urinary incontinence
* Voluntarily agreed to participate in the research

Exclusion Criteria:

* Benign prostatic hyperplasia
* Prostate cancer
* Congenital urinary anomalies
* Neurological or spinal cord injury,
* Diabetes mellitus
* Hypertension
* A mental disability
* Receive medical treatment for incontinence

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
A Change on Incontinence Severity Measured by The International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF) | 20 minutes before and 6 months after the training
  The primary outcome measure was the mean score change from baseline incontinence severity at 6 months measured by the International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF). The ICIQ-SF consists of a total of six items, including the birth date, gender and urinary incontinence characteristics. The score range of this scale is 0-21. High scores indicate increased urinary incontinence severity.

SECONDARY OUTCOMES:
The Urogenital Distress Inventory (UDI-6) | 20 minutes before and 6 months after the training
  UDI-6 is short forms of the scales developed by Uebersax et al. with six and seven questions, respectively. The Turkish validity study of these forms was made by Cam et al., who reported a Cronbach's alpha coefficient for UDI-6 as 0.74. In this study, the Cronbach's alpha coefficient for UDI-6 was 0.786 before training and 0.746 after the training implementations. Each item was scored between zero and 3, and the total score was calculated in the range of zero to 100. Higher scores obtained from these scales indicate that bladder function is worse.
The Incontinence Impact Questionnaire-7 (IIQ-7) | 20 minutes before and 6 months after the training
  IIQ-7 is short forms of the scales developed by Uebersax et al. with six and seven questions, respectively. The Turkish validity study of these forms was made by Cam et al., who reported a Cronbach's alpha coefficient for IIQ-7 as 0.87. In this study, the Cronbach's alpha coefficient for IIQ-7 was 0.933 before training and 0.902 after the training implementations. Each item was scored between zero and 3, and the total score was calculated in the range of zero to 100. Higher scores obtained from these scales indicate that bladder function is worse.

OTHER OUTCOMES:
The Urinary Incontinence Information Evaluation Form (UIIEF) | 20 minutes before and 6 months after the training
  Urinary Incontinence Information Evaluation Form (UIIEF) is an information form consisting of 10 multiple choice questions prepared by researchers literature-based and expert opinions. Each item is scored between 0-10 and the total score is calculated in the range of 0-100. The scores obtained from this form provide information about the change of information score means.

CONTACTS AND LOCATIONS:
Overall Officials: Hilal Tüzer, RN, PhD, Study Director — Ankara Yildirim Beyazıt University; Elif Gezginci, RN, PhD, Principal Investigator — Saglik Bilimleri Universitesi; Tuba Yılmazer, RN, PhD, Principal Investigator — Ankara Yildirim Beyazıt University
Locations (1):
- Ankara Yildirim Beyazit University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abrams P, Cardozo L, Fall M, Griffiths D, Rosier P, Ulmsten U, van Kerrebroeck P, Victor A, Wein A; Standardisation Sub-committee of the International Continence Society. The standardisation of terminology of lower urinary tract function: report from the Standardisation Sub-committee of the International Continence Society. Neurourol Urodyn. 2002;21(2):167-78. doi: 10.1002/nau.10052. No abstract available. PMID 11857671
- [Background] Stewart WF, Van Rooyen JB, Cundiff GW, Abrams P, Herzog AR, Corey R, Hunt TL, Wein AJ. Prevalence and burden of overactive bladder in the United States. World J Urol. 2003 May;20(6):327-36. doi: 10.1007/s00345-002-0301-4. Epub 2002 Nov 15. PMID 12811491
- [Background] Irwin DE, Milsom I, Hunskaar S, Reilly K, Kopp Z, Herschorn S, Coyne K, Kelleher C, Hampel C, Artibani W, Abrams P. Population-based survey of urinary incontinence, overactive bladder, and other lower urinary tract symptoms in five countries: results of the EPIC study. Eur Urol. 2006 Dec;50(6):1306-14; discussion 1314-5. doi: 10.1016/j.eururo.2006.09.019. Epub 2006 Oct 2. PMID 17049716
- [Background] Irwin DE, Abrams P, Milsom I, Kopp Z, Reilly K; EPIC Study Group. Understanding the elements of overactive bladder: questions raised by the EPIC study. BJU Int. 2008 Jun;101(11):1381-7. doi: 10.1111/j.1464-410X.2008.07573.x. Epub 2008 Mar 10. PMID 18336602
- [Background] Eapen RS, Radomski SB. Gender differences in overactive bladder. Can J Urol. 2016 Feb;23(Suppl 1):2-9. PMID 26924589
- [Background] Jeon E, Park HA. Development of the IMB Model and an Evidence-Based Diabetes Self-management Mobile Application. Healthc Inform Res. 2018 Apr;24(2):125-138. doi: 10.4258/hir.2018.24.2.125. Epub 2018 Apr 30. PMID 29770246
- [Background] Zarani F, Besharat MA, Sarami G, Sadeghian S. An information-motivation-behavioral skills (IMB) model-based intervention for CABG patients. Int J Behav Med. 2012 Dec;19(4):543-9. doi: 10.1007/s12529-011-9193-2. PMID 21948041
- [Background] Kiene SM, Fisher WA, Shuper PA, Cornman DH, Christie S, Macdonald S, Pillay S, Mahlase G, Fisher JD. Understanding HIV transmission risk behavior among HIV-infected South Africans receiving antiretroviral therapy: an information--motivation--behavioral skills model analysis. Health Psychol. 2013 Aug;32(8):860-8. doi: 10.1037/a0030554. Epub 2013 Mar 11. PMID 23477576
- [Background] Konkle-Parker DJ, Amico KR, McKinney VE. Effects of an intervention addressing information, motivation, and behavioral skills on HIV care adherence in a southern clinic cohort. AIDS Care. 2014;26(6):674-83. doi: 10.1080/09540121.2013.845283. Epub 2013 Oct 14. PMID 24116922
- [Background] Uebersax JS, Wyman JF, Shumaker SA, McClish DK, Fantl JA. Short forms to assess life quality and symptom distress for urinary incontinence in women: the Incontinence Impact Questionnaire and the Urogenital Distress Inventory. Continence Program for Women Research Group. Neurourol Urodyn. 1995;14(2):131-9. doi: 10.1002/nau.1930140206. PMID 7780440
- [Background] Cam C, Sakalli M, Ay P, Cam M, Karateke A. Validation of the short forms of the incontinence impact questionnaire (IIQ-7) and the urogenital distress inventory (UDI-6) in a Turkish population. Neurourol Urodyn. 2007;26(1):129-33. doi: 10.1002/nau.20292. PMID 17083117
- [Background] Aydin Sayilan A, Ozbas A. The Effect of Pelvic Floor Muscle Training On Incontinence Problems After Radical Prostatectomy. Am J Mens Health. 2018 Jul;12(4):1007-1015. doi: 10.1177/1557988318757242. Epub 2018 Mar 14. PMID 29540090
- [Background] Shell DF, Newman IM, Perry CM, Folsom AR. Changing intentions to use smokeless tobacco: an application of the IMB model. Am J Health Behav. 2011 Sep;35(5):568-80. doi: 10.5993/ajhb.35.5.6. PMID 22040618
- [Background] Walsh JL, Senn TE, Scott-Sheldon LA, Vanable PA, Carey MP. Predicting condom use using the Information-Motivation-Behavioral Skills (IMB) model: a multivariate latent growth curve analysis. Ann Behav Med. 2011 Oct;42(2):235-44. doi: 10.1007/s12160-011-9284-y. PMID 21638196
- [Background] Osborn CY, Egede LE. Validation of an Information-Motivation-Behavioral Skills model of diabetes self-care (IMB-DSC). Patient Educ Couns. 2010 Apr;79(1):49-54. doi: 10.1016/j.pec.2009.07.016. Epub 2009 Aug 21. PMID 19699601
- [Background] Mittal M, Senn TE, Carey MP. Intimate partner violence and condom use among women: does the information-motivation-behavioral skills model explain sexual risk behavior? AIDS Behav. 2012 May;16(4):1011-9. doi: 10.1007/s10461-011-9949-3. PMID 21484278
- [Background] Malow RM, Devieux JG, Stein JA, Rosenberg R, Lerner BG, Attonito J, Villalba K. Neurological function, information-motivation-behavioral skills factors, and risk behaviors among HIV-positive alcohol users. AIDS Behav. 2012 Nov;16(8):2297-308. doi: 10.1007/s10461-012-0246-6. PMID 22767030
- [Background] Ndebele M, Kasese-Hara M, Greyling M. Application of the information, motivation and behavioural skills model for targeting HIV risk behaviour amongst adolescent learners in South Africa. SAHARA J. 2012 Dec;9 Suppl 1:S37-47. doi: 10.1080/17290376.2012.744903. PMID 23234378
- [Background] Kudo Y. Effectiveness of a condom use educational program developed on the basis of the Information-Motivation-Behavioral Skills model. Jpn J Nurs Sci. 2013 Jun;10(1):24-40. doi: 10.1111/j.1742-7924.2012.00207.x. Epub 2012 Mar 30. PMID 23735087
- [Background] Ybarra ML, Korchmaros JD, Prescott TL, Birungi R. A Randomized Controlled Trial to Increase HIV Preventive Information, Motivation, and Behavioral Skills in Ugandan Adolescents. Ann Behav Med. 2015 Jun;49(3):473-85. doi: 10.1007/s12160-014-9673-0. PMID 25633626
- [Background] Ribeiro LH, Prota C, Gomes CM, de Bessa J Jr, Boldarine MP, Dall'Oglio MF, Bruschini H, Srougi M. Long-term effect of early postoperative pelvic floor biofeedback on continence in men undergoing radical prostatectomy: a prospective, randomized, controlled trial. J Urol. 2010 Sep;184(3):1034-9. doi: 10.1016/j.juro.2010.05.040. PMID 20643454
- [Background] Thuroff JW, Abrams P, Andersson KE, Artibani W, Chapple CR, Drake MJ, Hampel C, Neisius A, Schroder A, Tubaro A. EAU guidelines on urinary incontinence. Eur Urol. 2011 Mar;59(3):387-400. doi: 10.1016/j.eururo.2010.11.021. Epub 2010 Nov 24. PMID 21130559
- [Background] Nambiar AK, Bosch R, Cruz F, Lemack GE, Thiruchelvam N, Tubaro A, Bedretdinova DA, Ambuhl D, Farag F, Lombardo R, Schneider MP, Burkhard FC. EAU Guidelines on Assessment and Nonsurgical Management of Urinary Incontinence. Eur Urol. 2018 Apr;73(4):596-609. doi: 10.1016/j.eururo.2017.12.031. Epub 2018 Feb 3. PMID 29398262
- See also: Peyman N, Abdollahi M. Using of information-motivation-behavioral skills model on nutritional behaviors in controlling anemia among girl students. J Research&Health. 2016; 12 — http://www.k4health.org/sites/default/files/peyman_and_abdollahi_2016.pdf